CLINICAL TRIAL: NCT03082456
Title: Molecular Breast Imaging in Screening Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CMRPG2E0341
Record Dates: First submitted 2017-03-01; First posted 2017-03-17 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: molecular breast imaging; MBI; breast cancer; mammography; sonography; recall rate; diagnostic accuracy; breast echo; female population
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography; Ultrasonography, Mammary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Three breast screening modalities (Other): Subjects who have had mammography less than two years ago will receive MBI and breast ultrasound only. Other participants will receive three interventions including molecular breast imaging, mammography and breast ultrasound. The interval between each examination will be less than 6 months.
  Interventions: Diagnostic Test: Molecular breast imaging; Diagnostic Test: Mammography; Diagnostic Test: Breast ultrasound

INTERVENTIONS:
Diagnostic Test: Molecular breast imaging — Molecular breast imaging will be performed at 5-10 minutes after intravenous injection of 15-20 millicurie (mCi) Tc-99m sestamibi. Both craniocaudal (CC) view and mediolateral oblique (MLO) images of the breast are taken.
  Other Names: MBI
Diagnostic Test: Mammography — During the procedure, the breast is compressed using a dedicated mammography unit. Parallel-plate compression evens out the thickness of breast tissue to increase image quality by reducing the thickness of tissue that x-rays must penetrate, decreasing the amount of scattered radiation, reducing the required radiation dose, and holding the breast still (preventing motion blur). Both craniocaudal (CC) view and mediolateral oblique (MLO) images of the breast are taken.
  Other Names: Mammogram
Diagnostic Test: Breast ultrasound — Ultrasound investigation of breast is performed by members of breast cancer team. If abnormality is found by the procedure, biopsy will not be performed directly.
  Other Names: Breast sonography; Breast echo

SUMMARY:
The molecular breast imaging (MBI) is a potential modality to screen breast cancer. In this study, we compare and evaluate the recall rate/diagnostic efficiency of MBI, mammography and breast sonography, and aim to determine best ways of breast cancer screening.

DETAILED DESCRIPTION:
Keywords: molecular breast imaging, MBI, breast cancer, mammography, sonography

1. Background: In breast cancer screening, the sensitivity of mammography is about 71-96 %, but the sensitivity decreases in the three following groups: (1) under 50 years old; (2) dense breast parenchyma; (3) higher risk of breast cancer. The Health and Welfare Ministry data in recent 2 years showed Taiwanese women accepted mammography for screening in the ratio of only about 36%, representing many missed opportunities for early detection. One reason to reject mammography may be the discomfort caused by compression. To solve the above mammography possible weakness, other screening methods came into being, such as molecular breast imaging (MBI) of nuclear medicine. Radiotracer of Tc-99m sestamibi was found for targeting breast tumor 20 years ago, and approved by the FDA in 1997. However, the application is limited due to the suboptimal scanning camera design. Ten years later, the Mayo Clinics developed MBI technology, using small-sized semiconductor detectors. Then it become possible that the nuclear technologist have patient's breast tissue fit the detector in almost the same fashion of mammography without heavy compression.
2. Objective: The aim of this study is to evaluate the recall rate and diagnostic accuracy of MBI, mammography and breast echo, for female population.
3. Study design: Female patients referred to Nuclear Medicine Department for myocardial perfusion scan will be recruited in this study. It is because that MBI and myocardial perfusion scan share the same radiotracer. Then MBI will become additional scanning only. About 1800 female subjects will involve, and further mammography and/or breast sonography will be arranged within 6 months after MBI. Participants will be encouraged to receive mammography every 2 years and telephone survey. We hope that this study will help us to compare and evaluate the recall rate/diagnostic efficiency of MBI, mammography and breast sonography, and to determine best ways of breast cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* Female patients undergoing myocardial perfusion imaging will be eligible if they sign the informed consent.

Exclusion Criteria:

* They are unable to understand and sign the consent form
* They are physically unable to sit upright and still for 20 minutes.
* They have undergone breast surgery or breast biopsy within the last 12 months.
* They have had trauma to the breast tissue or undergone radiation treatment to the breast within the last 12 months.

Ages: 45 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Recall rate | 6 months
  The frequency with which a radiologist or physician interprets findings of an examination as positive

SECONDARY OUTCOMES:
Diagnostic efficacy | 6 months
  The sensitivity, specificity, positive predictive value and negative predictive value of each imaging modality

CONTACTS AND LOCATIONS:
Locations (1):
- TzuPei Su, Keelung, Taiwan

IPD SHARING:
Plan to Share IPD: No